CLINICAL TRIAL: NCT05389059
Title: The Value of Injectable Platelet Rich Fibrin With Volume Stable Collagen Matrix in Treatment of Multiple Gingival Recession; a Randomized Clinical Trial.
Brief Title: Injectable Platelet Rich Fibrin With Collagen Matrix in Treatment of Multiple Gingival Recession.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Basima Ghaffoori Ali, PHD student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 519622
Record Dates: First submitted 2022-04-24; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Gingival Diseases; Traumatic Injury
Keywords: Gingival Recession; Collagen Matrix; Plasma rich proten
MeSH Terms: conditions — Gingival Diseases; Wounds and Injuries; Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Other): Patients with Gingival recessions are type 1 recession RT1 (cairo et al,2011) which correspond to Miller I&II gingival recession.
  Interventions: Procedure: CAF+CM
- Experimental arm (Other): Patients with Gingival recessions are type 1 recession RT1 (cairo et al,2011) which correspond to Miller I&II gingival recession.
  Interventions: Procedure: CAF+CM; Procedure: I-PRF

INTERVENTIONS:
Procedure: CAF+CM — Periodontal surgery including CAF+CM application
Procedure: I-PRF — Periodontal surgery including CAF+CM application with i-PRF
  Arms: Experimental arm

SUMMARY:
This study is proposing the use of i-PRF clot as a scaffold for the XCM in order to obtain a novel biomaterial, incorporating active growth factors and collagen matrix in a single framework, based on the potential effect of i-PRF to enhance fibroblast activity and angiogenesis stimulation for treatment of multiple gingival recession.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least two localized gingival recessions on either sides of the maxilla and/or mandible excluding molar region.
* The cemento-enamel junction (CEJ) is visible in the teeth for root coverage procedures.
* All recessions are type 1recession RT1 (cairo et al,2011) which correspond to Miller I&II gingival recession
* All patients must demonstrate adequate plaque control with a fullmouth plaque score less than 20% and with .
* All patients at least 18 years of age and of both genders.

Exclusion Criteria:

* Smoker Patients .
* Patients with diabetes.
* Patients with a history of malignancy, radiotherapy, or chemotherapy for malignancy.
* pregnant or nursing women.
* Patients taking medications or having treatments with an effect on mucosal healing in general (e.g. steroids, large doses of antiinflammatory drugs).
* Patients with a disease affecting connective tissue metabolism.
* Patients allergic to collagen.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in gingival recession depth on the buccal sides of type one gingival recessionRT1 | Between the baseline preoperative measurement and follow-up at 3 months and 6 months
  The primary outcome of the study is the reduction in gingival recession depth on the buccal sides of RT1 gingival recession, between the baseline preoperative measurement and follow-up at 3 months and 6 months. The Recession Depth (RD) is Measured in millimeter (mm) from CEJ (Cemento-Enamel-Junction) to the gingival margin using UNC-15 probe.

SECONDARY OUTCOMES:
Improvement in Gingival Thickness (GT) | Between the baseline preoperative measurement and follow-up at 3 months and 6 months
  Gingival Thickness (GT) is determined at 1.5 mm apical to the gingival margin using a caliper (endodontic reamer#20) rounded to the nearest 0.1mm.
Improvement in the Keratinized Tissue Height (KTH) | Between the baseline preoperative measurement and follow-up at 3 months and 6 months
  Keratinized Tissue Height (KTH) is measured in millimeters (mm) taken at the mid buccal aspect of the involved teeth from the gingival margin to the muco-gingival junction, by a manual periodontal probe (UNC-15 probe,Hu-Friedy,Chicago,USA).
Reduction in the Recession Width (RW) | Between the baseline preoperative measurement and follow-up at 3 months and 6 months
  Recession Width (RW) is measured in millimeter (mm) at the Cement-Enamel Junction (CEJ) using UNC-15 probe.
Reduction in Probing Pocket Depth (PPD) | Between the baseline preoperative measurement and follow-up at 3 months and 6 months
  Probing Pocket Depth (PPD) is measured in millimeter (mm) from the gingival margin to the apical extend of the probe.
Reduction Clinical Attachment Level (CAL) | Between the baseline preoperative measurement and follow-up at 3 months and 6 months
  Clinical Attachment Level (CAL) is measured in millimeter (mm) from the CEJ to the apical extend of the probe.
Measuring Plaque-Index (PI) | Between the baseline preoperative measurement and follow-up at 3 months and 6 months
  Plaque-Index (PI) is measured as a percentage of the presence of Plaque on four surfaces of the teeth using a manual periodontal probe.
Measuring Bleeding On Probing (BOP) | Between the baseline preoperative measurement and follow-up at 3 months and 6 months
  Bleeding On Probing (BOP) is measured as a percentage of sites with bleeding on probing using a manual periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Basima Gh Ali, MSc, Principal Investigator — University of Baghdad; Thair AL Hassan, PHD, Study Director — University of Baghdad
Locations (1):
- University of Baghdad / College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No